CLINICAL TRIAL: NCT06524739
Title: Double-blind, Randomized, Placebo-controlled Phase 3 Study Evaluating Efficacy and Safety of IgPro20 (Subcutaneous Immunoglobulin, HIZENTRA®) in Post-COVID-19 Postural Orthostatic Tachycardia Syndrome (POTS)
Brief Title: Double-blind, Randomized, Placebo-controlled Study Evaluating Efficacy and Safety of IgPro20 in Post-COVID-19 POTS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision, not for safety reasons.
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IgPro20_3010; 2023-508744-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-26; First posted 2024-07-29 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Post-COVID Postural Orthostatic Tachycardia Syndrome
Keywords: POTS
MeSH Terms: interventions — Hizentra

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Period 1 (double-blind): Participant, Care Provider, Investigator, Outcomes Assessor
  Period 2 (open-label): No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IgPro20 (Experimental)
  Interventions: Biological: IgPro20
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: IgPro20 — IgPro20 is a 20% ready-to-use liquid formulation of polyvalent human immunoglobulin G (IgG) for subcutaneous (SC) administration
  Other Names: HIZENTRA®
  Arms: IgPro20
Biological: Placebo — 2% human albumin solution administered subcutaneously as a volume-matched dose to the experimental IMP.
  Arms: Placebo

SUMMARY:
This is a prospective, phase 3, multicenter, double-blind, randomized placebo-controlled study to investigate the efficacy, safety, and pharmacokinetics (PK) of repeat doses of IgPro20 in participants with post SARS-CoV-2 infection 2019 postural orthostatic tachycardia syndrome (post-Coronavirus Disease 2019 [COVID-19] POTS [post-COVID-POTS]).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent and be willing and, in the opinion of the investigator, able to adhere to all protocol requirements.
2. Males and females aged ≥ 18 at the time of providing written informed consent.
3. Diagnosis of post-COVID POTS, defined by both a preceding COVID-19 infection based on confirmed historical documentation and onset of POTS symptoms developing within 4 months after COVID-19 infection as defined per consensus criteria.
4. COMPASS-31 score of at least 40 at the Screening visit.
5. Positive confirmatory standardized standing test (ie, HR increase of ≥ 30 bpm [≥ 40 bpm for participants aged 18 to 19 years] within 10 minutes in the absence of orthostatic hypotension) at the Screening visit.

Exclusion Criteria:

1. Treatment with Immunoglobulin G (IgG) or plasmapheresis within 12 weeks before Screening
2. Symptoms and / or diagnosis of or receiving treatment for POTS before COVID-19 infection
3. Prior diagnosis of or receiving current treatment at Screening for the following conditions (unless onset was related to the inciting POTS-associated COVID-19 infection): certain neurologic, autoimmune, endocrine, cardiac, or other disorders, and pre-existing psychiatric disorders
4. Presence of active infections, including human immunodeficiency virus infection, hepatitis B, hepatitis C, active SARS-CoV-2 infection, or any uncontrolled systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Proportion of participants no longer meeting diagnostic criteria of post-COVID POTS as measured by standardized standing test (ie, no longer experiencing HR increase of ≥ 30 bpm, in the absence of 20 mmHg decrease of SBP [orthostatic hypotension]) | At screening, and at week 25

SECONDARY OUTCOMES:
Change from baseline in orthostatic intolerance score of COMPASS-31 | At baseline and at week 25
  The Composite Autonomic Symptom Score 31 (COMPASS-31) is a self-reported questionnaire that measures autonomic symptoms related to 6 domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder and pupillomotor. The treatment effect of interest is differences from baseline in the orthostatic intolerance score of COMPASS-31.
Change from baseline in COMPASS-31 total score | At baseline and at week 25
  The COMPASS-31 is a self-reported questionnaire that measures autonomic symptoms related to 6 domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder and pupillomotor. This questionnaire generates a weighted score from 0 to 100, with higher scores representing higher symptom burden.
Change from baseline in heart rate increase within 10 minutes of standing test | At baseline and at Week 25
Number of participants with treatment-emergent adverse events (TEAEs), related TEAEs, serious TEAEs and related serious TEAEs | After treatment, for up to 57 weeks
Percentage of participants with TEAEs, related TEAEs, serious TEAEs and related serious TEAEs | After treatment, for up to 57 weeks
Number of participants with electrocardiogram (ECG) abnormalities | At baseline, at Week 25 and at Week 53
Percentage of participants with ECG abnormalities | At baseline, at Week 25 and at Week 53
Change from baseline in ECG abnormalities | At baseline, at Week 25 and at Week 53

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (38):
- United States (34):
  - University of Alabama Hospital at Birmingham, Birmingham, Alabama
  - Center for Complex Neurology, EDS & POTS, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Arkansas Cardiology Clinic - Little Rock, Little Rock, Arkansas
  - UC San Diego Health, La Jolla, California
  - University of california Irvine, Orange, California
  - National Jewish Health, Denver, Colorado
  - Hope Research Network, Miami, Florida
  - Well Pharma Medical Research, Corp, Miami, Florida
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Velocity Clinical Research, Metairie, New Orleans, Louisiana
  - Johns Hopkins Bayview Medical Center PMR, Baltimore, Maryland
  - Mass General Brigham (Massachusetts General Hospital), Belmont, Massachusetts
  - Profound Research LLC at Millennium Affiliated Physicians, Farmington Hills, Michigan
  - Velocity Clinical Research - Lincoln, Lincoln, Nebraska
  - Dysautonomia Clinic, Buffalo, New York
  - NYU Langone Health South Shore Neurologic Associates, Patchogue, New York
  - Duke University Medical Center, Durham, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Velocity Clinical Research - Union, Union, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Austin Dell Medical School, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Sunbeam Clinical Research, McKinney, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Bateman Horne Center, Salt Lake City, Utah
  - Metrodora Institute, West Valley City, Utah
  - Velocity Clinical Research - Hampton, Hampton, Virginia
  - VCU Health, Richmond, Virginia
- Canada (4):
  - Libin Cardiovascular Institute University of Calgary, Calgary
  - University of Alberta Hospital, Edmonton
  - McGill University Health Centre, Québec
  - Ciussse-Chus, Sherbrooke

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.